CLINICAL TRIAL: NCT06925113
Title: A Retrospective, Non-interventional, Multicenter Study to Investigate the Prevalence of HER2 IHC 3+ and Characterize the Clinicopathologic Features of Gynecologic Cancers in Taiwan -The HERGYN Study
Brief Title: A Study to Investigate the Prevalence of Human Epidermal Growth Factor Receptor 2 (HER2) Immunohistochemistry (IHC) 3+ and Characterize the Clinicopathologic Features of Gynecologic Cancers in Taiwan
Acronym: HERGYN
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS8201-TWMA-Gyn-4001
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancers; Endometrial Cancer; Ovarian Cancer
Keywords: gynecology; HER2 IHC; prevalence; Taiwan; retrospective
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recurrent or advanced gynecologic cancers: Recurrent or advanced endometrial cancer, ovarian cancer, or cervical cancer diagnosed between 2022 to 2024

SUMMARY:
Trastuzumab Deruxtecan (T-DXd) is a humanized anti-HER2 monoclonal antibody covalently linked to DXd, which is a topoisomerase 1 inhibitor. T-DXd has been approved for the treatment of HER2-positive breast cancer, HER2-mutated lung cancer, HER2-positive gastric cancer, and HER2-low breast cancer in Taiwan. Aside from clinical benefits in the above cancers, the DESTINY-PanTumor02 (NCT04482309) Phase II trial showed that T-DXd continued to demonstrate clinically meaningful and durable responses and survival benefits in previously treated patients across multiple HER2-expressing advanced solid tumors.

Among multiple types of solid tumors in the DESTINY-PanTumor02 trial, T-DXd showed a high confirmed objective response rate in heavily treated HER2 IHC 3+ endometrial cancer (EC, 84.6%, 11/13), ovarian cancer (OC, 63.6%, 7/11), and cervical cancer (CC, 75%, 6/8).

Previous evidence showed that HER2-expressing gynecologic cancers have limited treatment options and have poor prognoses under standard therapies. Data from DESTINY-PanTumor02 therefore serve as supporting evidence for T-DXd to become a potential therapeutic option for these HER2-expressing gynecologic cancers.

In August 2023, T-DXd received the FDA-designated breakthrough therapy designations and was approved in April 2024 for treating unresectable and metastatic HER2 IHC 3+ solid tumors that have progressed after prior treatment or lack satisfactory alternative options. The National Comprehensive Cancer Network (NCCN) has included T-DXd as a treatment option for HER2-positive endometrial, ovarian, and cervical carcinomas in their guidelines as of V1 2024.

However, the prevalence rate of HER2 IHC 3+ in recurrent advanced endometrial, ovarian, and cervical cancers in Taiwan remains unclear. Limited information is available regarding the HER2 amplification rate by ISH for specific cancer types.

In this retrospective, non-interventional study, the investigators aim to explore the prevalence of HER2 IHC 3+ in recurrent advanced endometrial, ovarian, and cervical cancers in Taiwan. The clinicopathologic characteristics will also be described, using information abstracted from the medical charts, to better understand and characterize the patient profiles of recurrent advanced endometrial, ovarian, and cervical cancers in Taiwan.

DETAILED DESCRIPTION:
It is a non-interventional, multicenter, retrospective study to investigate the prevalence rate of HER2 IHC 3+ determined by IHC and characterize the clinicopathologic features of recurrent advanced endometrial, ovarian, and cervical cancers in Taiwan. The study plans to include approximately 170 patients with endometrial cancer, 170 patients with ovarian cancer, and 170 patients with cervical cancer from five hospitals in Taiwan.

The study will retrospectively review medical charts to screen potential patients for enrollment in the study. A pathologist investigator meeting aligned with ASCO/CAP guidelines for scoring HER2 in Gastroesophageal Adenocarcinoma will be held to ensure the concordance of IHC scoring among different sites before patient enrollment.

Once enrolled, the study will collect the most recent and qualified archived tissue samples from recurrent advanced tumors of eligible patients to perform HER2 IHC test using Ventana 4B5 assay by pathologists per standard operational procedures at each hospital (after pathologist investigator meeting). If the patient already had HER2 IHC slides stained with Ventana 4B5 assay from recurrent advanced tumors, the pathologist will rescore the HER2 IHC data without conducting HER2 IHC staining again.

For patients who have archived primary tumor tissue samples before recurrence (2024 or before, regardless of FIGO stage), the study will also collect the primary tumor tissue samples before recurrence, which are qualified and sufficient for performing HER2 IHC test using Ventana 4B5 assay by pathologists per standard operational procedures at each hospital to analyze the changes in HER2 status after recurrence. If the patient already had HER2 IHC slides stained with Ventana 4B5 assay from the primary tumors before recurrence, the pathologist will rescore the HER2 IHC data without conducting HER2 IHC staining again.

In addition to the HER2 IHC test, patient-level data, including demographics, clinicopathologic characteristics, standard and exploratory diagnostic information (e.g., histopathology and biomarkers), and the clinical presentation of gynecologic cancers (e.g., FIGO stage, metastatic sites, etc.) will be abstracted from medical charts of enrolled patients after de-identification.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 years when their clinical data are reviewed
2. Patients who fulfill ONE of the following criteria

   * Imaging or histological diagnosis of recurrent advanced endometrial cancer during 2022 to 2024, AND have tissue samples from recurrent advanced tumor (regardless of lines of received treatment) during 2022 to 2024 for HER2 IHC test (most recent and qualified pre-enrollment tumor sample must be provided)
   * Imaging or histological diagnosis of recurrent advanced ovarian cancer during 2022 to 2024, AND have tissue samples from recurrent advanced tumor (regardless of lines of received treatment) during 2022 to 2024 for HER2 IHC test (most recent and qualified pre-enrollment tumor sample must be provided)
   * Imaging or histological diagnosis of recurrent advanced cervical cancer during 2022 to 2024, AND have tissue samples from recurrent advanced tumor (regardless of lines of received treatment) during 2022 to 2024 for HER2 IHC test (most recent and qualified pre-enrollment tumor sample must be provided)

Exclusion Criteria:

1. Without FFPE tumor sample from recurrent advanced tumors (specimens with limited tumor content and fine needle aspirates are inadequate for defining tumor HER2 status)
2. With the retrospective nature and the use of anonymous clinical data, IRB/IEC/EC may grant permission to waive informed consent in this study. If the informed consent is not waived, patients or representatives who are not willing to provide written informed consent cannot be enrolled.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Recurrent or advanced endometrial cancer, ovarian cancer, or cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
To understand the prevalence rate of HER2 IHC 3+ in recurrent advanced endometrial cancer, ovarian cancer, and cervical cancer in Taiwan | from Jan 2022 to Dec 2024

SECONDARY OUTCOMES:
To understand the prevalence rate of HER2 IHC 2+, 1+, and 0 in recurrent advanced endometrial cancer, ovarian cancer, and cervical cancer in Taiwan | from Jan 2022 to Dec 2024

OTHER OUTCOMES:
To assess changes in HER2 IHC score between primary tumor before recurrence and recurrent advanced tumor | from Jan 2022 to Dec 2024
  To assess changes in HER2 IHC score between primary tumor before recurrence and recurrent advanced tumor by calculating the changes in HER2 IHC score (HER2 IHC score is categorized into 0, 1+, 2+, and 3+)
To assess the correlation between HER2 IHC status and other biomarkers in gynecologic cancers by correlation coefficient analysis | from Jan 2022 to Dec 2024

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/